CLINICAL TRIAL: NCT04809220
Title: A Randomized, Double-Blind, Parallel Arm Study of the Efficacy and Safety of Two Doses of Dulaglutide in Combination With a Single Oral Antihyperglycemic Medication or as Monotherapy in Japanese Patients With Type 2 Diabetes Mellitus (AWARD-JPN: Assessment of Weekly Administration of LY2189265 in Diabetes - JAPAN)
Brief Title: A Study of Two Doses of Dulaglutide (LY2189265) in Japanese Patients With Type 2 Diabetes
Acronym: AWARD-JPN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17779; H9X-JE-GBGQ (Other: Eli Lilly and Company)
Record Dates: First submitted 2021-03-19; First posted 2021-03-22 (Actual); Results first posted 2023-09-21 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-04

CONDITIONS: Diabetes Mellitus; Diabetes Mellitus, Type 2; Glucose Metabolism Disorders; Metabolic Disease; Endocrine System Diseases; Hypoglycemic Agents; Type 2 Diabetes Mellitus (T2DM)
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2; Glucose Metabolism Disorders; Metabolic Diseases; Endocrine System Diseases | interventions — dulaglutide; Hypoglycemic Agents

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Dulaglutide 1.5 milligram (mg) (Experimental): Participants received 1.5 mg of dulaglutide given weekly subcutaneously (SC) during the 52-week treatment period. Dulaglutide will be given alone or in combination with 1 oral antihyperglycemic medication (OAM). Participants on dipeptidyl peptidase-4 inhibitors (DPP-4i) discontinued DPP-4i at randomization and was regarded as monotherapy of dulaglutide, other OAMs continued at same dose during study period and were regarded as combination therapy with dulaglutide.
  Interventions: Drug: Dulaglutide; Drug: Oral antihyperglycemics
- Dulaglutide 0.75 mg (Active Comparator): Participants received 0.75 mg of dulaglutide given weekly SC during the 52-week treatment period. Dulaglutide will be given alone or in combination with 1 OAM. Participants on DPP-4i discontinued DPP-4i at randomization and was regarded as monotherapy of dulaglutide, other OAMs continued at same dose during study period and were regarded as combination therapy with dulaglutide.
  Interventions: Drug: Dulaglutide; Drug: Oral antihyperglycemics

INTERVENTIONS:
Drug: Dulaglutide — Administered SC
  Other Names: LY2189265
Drug: Oral antihyperglycemics — Administered orally

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of 2 doses of dulaglutide in Japanese participants with type 2 diabetes. The study duration is approximately 58 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Participants with type 2 diabetes (T2D) ≥ 6 months according to the World Health Organization (WHO) classification.
* Treated with stable doses of a single OAM for at least 8 weeks prior to screening; the dose must be more than or equal to minimum maintenance dose.
* Have the following HbA1c result at screening.

  * Participants taking DPP-4i: ≥7.5% and ≤9.5%,
  * Participants taking another OAM: ≥8.0% and ≤10.0%
* Stable body weight for at least 8 weeks prior to screening or not changed by more than 5 % in the past 8 weeks
* Have a body mass index (BMI) ≥18.5 kilogram/square meter (kg/m²) and <35 kg/m² at Day 1.

Exclusion Criteria:

* Have type 1 diabetes (T1D)
* Have a history of ≥1 episode of ketoacidosis or hyperosmolar state/coma
* Have had any myocardial infarction (MI), heart failure or cerebrovascular accident (stroke)
* Have a known clinically significant gastric empty abnormality
* Have acute or chronic hepatitis
* Have had chronic or acute pancreatitis
* Have any self or family history of type 2A or type 2B multiple endocrine neoplasia in the absence of known C-cell hyperplasia
* Have any self or family history of medullary C-cell hyperplasia, focal hyperplasia, or carcinoma (including sporadic, familial, or part of Multiple endocrine neoplasia (MEN) 2A or 2B syndrome)
* Have evidence of significant, active autoimmune abnormality
* Have evidence of significant, uncontrolled endocrine abnormality
* Have active or untreated malignancy, or have been in remission from clinically significant malignancy (other than basal cell or squamous cell skin cancer) for less than 5 years
* Have any hematologic condition that may interfere with HbA1c measurement

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 591 (Actual)
Dates: Start 2021-04-13 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2023-04-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon- Fri 9 AM- 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (44):
- Japan (44):
  - Nakayama Clinic, Nagoya, Aichi-ken
  - Tosaki Clinic for Diabetes and Endocrinology, Nagoya, Aichi-ken
  - Kashiwa City Hospital, Kashiwa, Chiba
  - Kobari General Clinic, Noda, Chiba
  - Nippon Kokan Fukuyama Hospital, Fukuyama-shi, Hiroshima
  - Yamagata Naika Clinic, Asahikawa, Hokkaido
  - Hasegawa Medical Clinic, Chitose, Hokkaido
  - Yuri Ono Clinic, Sapporo, Hokkaido
  - Manda Memorial Hospital, Sapporo, Hokkaido
  - Miyanosawa Clinic of Internal Medicine and Cardiology, Sapporo, Hokkaido
  - Takabe Diabetes Clinic, Himeji, Hyōgo
  - Nakamoto Internal Medicine Clinic, Mito, Ibaraki
  - Nakakinen clinic, Naka, Ibaraki
  - Nishiyamadou Keiwa Hospital, Naka, Ibaraki
  - Hayashi Diabetes Internal Medicine Clinic, Chigasaki, Kanagawa
  - Shonan Takai Clinic, Kamakura, Kanagawa
  - Takai Internal Medicine Clinic, Kamakura-shi, Kanagawa
  - Yamagishi Clinic Sagamiono, Sagamihara, Kanagawa
  - Medical Corporation Yuga Tsuruma Kaneshiro Diabetes Clinic, Yamato-shi, Kanagawa
  - Seiryo Internal Medicine, Iwanuma, Miyagi
  - Gibo Hepatology Clinic, Matsumoto, Nagano
  - Shiraiwa Medical Clinic, Kashihara, Osaka
  - Medical Corporation Heishinkai OCROM Clinic, Suita-shi, Osaka
  - Sugiura Internal Medicine Clinic, Sōka, Saitama
  - Seiwa Clinic, Adachi-ku, Tokyo
  - Tokyo-Eki Center-building Clinic, Chuo-ku, Tokyo
  - Medical Corporation Chiseikai Tokyo Center Clinic, Chuo-ku, Tokyo
  - Fukuwa Clinic, Chuo-ku, Tokyo
  - Hachioji Diabetes Clinic, Hachiōji, Tokyo
  - Minamino Cardiovascular Hospital, Hachiōji, Tokyo
  - Yutenji Medical Clinic, Meguro-ku, Tokyo
  - Kanno Naika, Mitaka, Tokyo
  - Heishinkai Medical Group ToCROM Clinic, Shinjuku-ku, Tokyo
  - Nomura Clinic, tabashi City, Tokyo
  - Futata Tetsuhiro Clinic, Fukuoka
  - Yoshimura Clinic, Kumamoto
  - Jinnouchi Hospital, Kumamoto
  - Heiwadai Hospital, Miyazaki
  - Ota Diabetes Internal Medicine Clinic, Nagano
  - AMC Nishiumeda Clinic, Osaka
  - Kitada Clinic, Osaka
  - Osaka Metropolitan Univ Hosp, Osaka
  - Nanko Clinic, Osaka
  - Abe Clinic, Ōita

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 591 participants were randomized in the study. However, due to good clinical practice (GCP) compliance issues identified at one of the investigative sites, all 5 participants from that site were excluded from the study analyses.
Groups:
- Dulaglutide 1.5 Milligram (mg): Participants received 1.5 mg of dulaglutide given weekly SC during the 52-week treatment period. Dulaglutide will be given alone or in combination with 1 OAM. Participants on DPP-4i discontinued DPP-4i at randomization and was regarded as monotherapy of dulaglutide, other OAMs continued at same dose during study period and were regarded as combination therapy with dulaglutide.
Period: Overall Study
Arm/Group | Dulaglutide 1.5 Milligram (mg) | Dulaglutide 0.75 mg
Started | 395 | 196
Exposed to at Least 1 Dose of Study Intervention (Excluding the GCP Compliance Investigative Site) | 391 | 195
Completed | 377 | 190
Not Completed | 18 | 6
Not completed — Adverse Event | 4 | 0
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 3 | 0
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 9 | 5
Not completed — Due to long-term overseas business trips | 1 | 0

BASELINE CHARACTERISTICS:
Population: All randomly assigned participants, excluding the GCP compliance investigative site, who were exposed to at least 1 dose of study intervention.
Groups:
- Dulaglutide 1.5 mg: Participants received 1.5 mg of dulaglutide given weekly SC during the 52-week treatment period. Dulaglutide will be given alone or in combination with 1 OAM. Participants on DPP-4i discontinued DPP-4i at randomization and was regarded as monotherapy of dulaglutide, other OAMs continued at same dose during study period and were regarded as combination therapy with dulaglutide.
- Total: Total of all reporting groups
Arm/Group | Dulaglutide 1.5 mg | Dulaglutide 0.75 mg | Total
Number analyzed (Participants) | 391 | 195 | 586
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.10 (10.70) | 60.70 (10.74) | 60.30 (10.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 113 | 53 | 166
  Male | 278 | 142 | 420
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 391 | 195 | 586
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 391 | 195 | 586
Hemoglobin A1c (HbA1c) [Mean (Standard Deviation); unit: Percentage of HbA1c] — HbA1c is the glycosylated fraction of hemoglobin A. It is measured to identify average plasma glucose concentration over prolonged periods of time.
  Percentage of HbA1c | 8.61 (0.62) | 8.61 (0.60) | 8.61 (0.61)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin A1c (HbA1c) at Week 26
Description: HbA1c is the glycosylated fraction of hemoglobin A. It is measured to identify average plasma glucose concentration over prolonged periods of time. Least Squares (LS) mean was determined by mixed model repeated measures (MMRM) model with Baseline + Pre-study oral antihyperglycemic medication (OAM) Group 1 + Treatment + Time + Treatment × Time as variables.
Time Frame: Baseline, Week 26
Population: All randomly assigned participants, excluding the GCP compliance investigative site, who were exposed to at least 1 dose of study intervention and had at least one post baseline value for this analysis.
Measure: Least Squares Mean (Standard Error); unit: Percentage of HbA1c
Arm/Group | Dulaglutide 1.5 mg | Dulaglutide 0.75 mg
Number analyzed (Participants) | 383 | 193
Percentage of HbA1c | -1.53 (0.043) | -1.25 (0.060)
Statistical Analysis 1: Comparison: Dulaglutide 1.5 mg vs Dulaglutide 0.75 mg; Test type: Superiority; p < .001, Mixed Models Analysis; LS Mean Difference = -0.29, 95% CI 2-sided [-0.43 to -0.14]

2. Secondary Outcome: Change From Baseline in HbA1c at Week 52
Description: HbA1c is the glycosylated fraction of hemoglobin A. It is measured to identify average plasma glucose concentration over prolonged periods of time. LS mean was determined by MMRM model with Baseline + Pre-study OAM Group 1 + Treatment + Time + Treatment × Time as variables.
Time Frame: Baseline, Week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percentage of HbA1c
Arm/Group | Dulaglutide 1.5 mg | Dulaglutide 0.75 mg
Number analyzed (Participants) | 383 | 193
Percentage of HbA1c | -1.50 (0.046) | -1.19 (0.065)
Statistical Analysis 1: Comparison: Dulaglutide 1.5 mg vs Dulaglutide 0.75 mg; Test type: Superiority; p < .001, Mixed Models Analysis; LS Mean Difference = -0.31, 95% CI 2-sided [-0.47 to -0.15]

3. Secondary Outcome: Percentage of Participants Achieving HbA1c Target ≤6.5% and <7.0%
Description: HbA1c is the glycosylated fraction of hemoglobin A. It is measured to identify average plasma glucose concentration over prolonged periods of time. The odds ratios, confidence intervals, and p-values were determined by generalized linear mixed model (GLM) with Baseline + Pre-study OAM Group 1 + Treatment + Time + Treatment × Time as variables.
Time Frame: Week 52
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Dulaglutide 1.5 mg | Dulaglutide 0.75 mg
Number analyzed (Participants) | 354 | 174
Percentage of participants
  HbA1c ≤ 6.5% | 22.88 | 21.26
  HbA1c < 7% | 46.33 | 38.51
Statistical Analysis 1: Comparison: Dulaglutide 1.5 mg vs Dulaglutide 0.75 mg; For HbA1c ≤6.5%; Test type: Superiority; p = 0.560, Generalized Linear Mixed Model (GLM); Odds Ratio (OR) = 1.15, 95% CI 2-sided [0.71 to 1.87]
Statistical Analysis 2: Comparison: Dulaglutide 1.5 mg vs Dulaglutide 0.75 mg; For HbA1c < 7%; Test type: Superiority; p = 0.028, Generalized Linear Mixed Model (GLM); Odds Ratio (OR) = 1.61, 95% CI 2-sided [1.05 to 2.45]

4. Secondary Outcome: Change From Baseline in Fasting Serum Glucose (FSG)
Description: FSG is a test to determine sugar levels in serum sample after an overnight fast. LS mean was determined by MMRM model with Baseline + Baseline HbA1c (High, Low) Group, OAM-based + Pre-study OAM Group 1 + Treatment + Time + Treatment*Time as variables.
Time Frame: Baseline, Week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: milligrams per deciliter (mg/dL)
Arm/Group | Dulaglutide 1.5 mg | Dulaglutide 0.75 mg
Number analyzed (Participants) | 382 | 191
milligrams per deciliter (mg/dL) | -42.4 (1.47) | -33.1 (2.09)
Statistical Analysis 1: Comparison: Dulaglutide 1.5 mg vs Dulaglutide 0.75 mg; Test type: Superiority; p < .001, Mixed Models Analysis; LS Mean Difference = -9.4, 95% CI 2-sided [-14.4 to -4.3]

5. Secondary Outcome: Change From Baseline in 6-point Self-Monitored Blood Glucose (SMBG)
Description: SMBG 6-point profiles were measured at morning (premeal-fasting, 2-hour post meal), midday (premeal, 2-hour post meal), and evening (premeal, 2-hour post meal). LS mean was determined by analysis of covariance (ANCOVA) model with Baseline + Baseline HbA1c (High, Low) Group, OAM-based + Pre-study OAM Group 1 + Treatment as variables.
Time Frame: Baseline, Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Dulaglutide 1.5 mg | Dulaglutide 0.75 mg
Number analyzed (Participants) | 362 | 185
mg/dL
  Morning premeal-fasting | -45.6 (1.33) | -38.4 (1.86)
  Morning 2-hour post meal: number analyzed (Participants) | 361 | 184
  Morning 2-hour post meal | -70.6 (2.42) | -60.5 (3.39)
  Midday premeal: number analyzed (Participants) | 361 | 185
  Midday premeal | -55.3 (1.77) | -47.0 (2.47)
  Midday 2-hour post meal: number analyzed (Participants) | 361 | 184
  Midday 2-hour post meal | -73.7 (2.37) | -61.2 (3.32)
  Evening premeal | -50.3 (1.60) | -46.4 (2.24)
  Evening 2-hour post meal: number analyzed (Participants) | 360 | 184
  Evening 2-hour post meal | -61.1 (2.27) | -49.8 (3.18)
Statistical Analysis 1: Comparison: Dulaglutide 1.5 mg vs Dulaglutide 0.75 mg; Morning premeal-fasting; Test type: Superiority; p = 0.002, ANCOVA; LS Mean Difference = -7.2, 95% CI 2-sided [-11.7 to -2.7]
Statistical Analysis 2: Comparison: Dulaglutide 1.5 mg vs Dulaglutide 0.75 mg; Morning 2-hour post meal; Test type: Superiority; p = 0.016, ANCOVA; LS Mean Difference = -10.1, 95% CI 2-sided [-18.3 to -1.9]
Statistical Analysis 3: Comparison: Dulaglutide 1.5 mg vs Dulaglutide 0.75 mg; Midday premeal; Test type: Superiority; p = 0.007, ANCOVA; LS Mean Difference = -8.3, 95% CI 2-sided [-14.2 to -2.3]
Statistical Analysis 4: Comparison: Dulaglutide 1.5 mg vs Dulaglutide 0.75 mg; Midday 2-hour post meal; Test type: Superiority; p = 0.002, ANCOVA; LS Mean Difference = -12.5, 95% CI 2-sided [-20.5 to -4.5]
Statistical Analysis 5: Comparison: Dulaglutide 1.5 mg vs Dulaglutide 0.75 mg; Evening premeal; Test type: Superiority; p = 0.158, ANCOVA; LS Mean Difference = -3.9, 95% CI 2-sided [-9.3 to 1.5]
Statistical Analysis 6: Comparison: Dulaglutide 1.5 mg vs Dulaglutide 0.75 mg; Evening 2-hour post meal; Test type: Superiority; p = 0.004, ANCOVA; LS Mean Difference = -11.3, 95% CI 2-sided [-19.0 to -3.7]

6. Secondary Outcome: Change From Baseline in Body Weight
Description: LS mean was determined by MMRM model with Baseline + Baseline HbA1c (High, Low) Group, OAM-based + Pre-study OAM Group 1 + Treatment + Time + Treatment*Time as variables.
Time Frame: Baseline, Week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: kilogram (kg)
Arm/Group | Dulaglutide 1.5 mg | Dulaglutide 0.75 mg
Number analyzed (Participants) | 383 | 193
kilogram (kg) | -0.5 (0.14) | -0.2 (0.19)
Statistical Analysis 1: Comparison: Dulaglutide 1.5 mg vs Dulaglutide 0.75 mg; Test type: Superiority; p = 0.213, Mixed Models Analysis; LS Mean Difference = -0.3, 95% CI 2-sided [-0.8 to 0.2]

ADVERSE EVENTS:
Time Frame: Baseline to Week 56.
Description: All randomly assigned participants, excluding the GCP compliance investigative site, who were exposed to at least 1 dose of study intervention. Gender specific events only occurring in male or female participants have had the number of participants At Risk adjusted accordingly.
Arm/Group | Dulaglutide 1.5 mg | Dulaglutide 0.75 mg
All-Cause Mortality (participants affected / at risk) | 1/391 | 0/195
Serious Adverse Events (participants affected / at risk) | 15/391 | 7/195
Other Adverse Events (participants affected / at risk) | 298/391 | 143/195
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Dulaglutide 1.5 mg (N=391) | Dulaglutide 0.75 mg (N=195)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Retinal haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Vitreous haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
Covid-19 (Infections and infestations) | 1 (1) | 0 (0)
Covid-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cervix carcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/113 (1) | 0/53 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Brain stem haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Lateral medullary syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Dulaglutide 1.5 mg (N=391) | Dulaglutide 0.75 mg (N=195)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Splenomegaly (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 2 (2)
Arteriosclerosis coronary artery (Cardiac disorders) | 2 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Bundle branch block right (Cardiac disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 2 (2) | 3 (4)
Supraventricular extrasystoles (Cardiac disorders) | 1 (1) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 2 (2) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Deafness neurosensory (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Presbyacusis (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Sudden hearing loss (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 3 (3) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 2 (2)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Age-related macular degeneration (Eye disorders) | 1 (1) | 0 (0)
Asthenopia (Eye disorders) | 2 (2) | 2 (2)
Blepharitis (Eye disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 7 (7) | 2 (2)
Central serous chorioretinopathy (Eye disorders) | 1 (1) | 0 (0)
Conjunctival deposit (Eye disorders) | 1 (1) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 1 (1) | 0 (0)
Corneal disorder (Eye disorders) | 1 (1) | 0 (0)
Diabetic retinal oedema (Eye disorders) | 0 (0) | 1 (1)
Diabetic retinopathy (Eye disorders) | 7 (7) | 2 (2)
Dry eye (Eye disorders) | 3 (4) | 1 (1)
Eczema eyelids (Eye disorders) | 0 (0) | 1 (1)
Glaucoma (Eye disorders) | 2 (2) | 1 (1)
Macular oedema (Eye disorders) | 0 (0) | 1 (1)
Ocular hyperaemia (Eye disorders) | 1 (1) | 0 (0)
Ocular hypertension (Eye disorders) | 1 (1) | 0 (0)
Retinal haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Retinal tear (Eye disorders) | 1 (1) | 0 (0)
Retinal vein occlusion (Eye disorders) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 24 (26) | 5 (5)
Abdominal distension (Gastrointestinal disorders) | 8 (8) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (3)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 2 (2)
Anal fissure haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chronic gastritis (Gastrointestinal disorders) | 4 (4) | 6 (6)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 49 (51) | 17 (17)
Dental caries (Gastrointestinal disorders) | 3 (3) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 40 (138) | 16 (17)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 14 (17) | 6 (6)
Ectopic gastric mucosa (Gastrointestinal disorders) | 1 (1) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Eructation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Faeces hard (Gastrointestinal disorders) | 1 (1) | 0 (0)
Faeces soft (Gastrointestinal disorders) | 3 (3) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric disorder (Gastrointestinal disorders) | 3 (4) | 0 (0)
Gastric polyps (Gastrointestinal disorders) | 4 (4) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastritis erosive (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 2 (3) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 10 (10) | 2 (2)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 1 (2)
Gingival pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 2 (2)
Melaena (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 35 (66) | 9 (9)
Pancreatic cyst (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatic duct dilatation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Periodontal disease (Gastrointestinal disorders) | 3 (3) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 4 (4) | 0 (0)
Toothache (Gastrointestinal disorders) | 3 (3) | 3 (3)
Vomiting (Gastrointestinal disorders) | 11 (23) | 2 (2)
Application site pruritus (General disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 2 (2) | 3 (5)
Chills (General disorders) | 0 (0) | 2 (2)
Cyst (General disorders) | 1 (1) | 0 (0)
Discomfort (General disorders) | 1 (1) | 0 (0)
Face oedema (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 2 (3)
Feeling abnormal (General disorders) | 1 (1) | 0 (0)
Injection site bruising (General disorders) | 2 (2) | 2 (6)
Injection site erythema (General disorders) | 1 (1) | 3 (3)
Injection site induration (General disorders) | 0 (0) | 1 (1)
Injection site pain (General disorders) | 1 (1) | 3 (3)
Injection site pruritus (General disorders) | 5 (27) | 2 (2)
Injection site reaction (General disorders) | 11 (52) | 5 (58)
Injection site swelling (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 14 (14) | 5 (7)
Pyrexia (General disorders) | 39 (48) | 14 (19)
Thirst (General disorders) | 1 (1) | 0 (0)
Vaccination site pain (General disorders) | 3 (3) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0)
Gallbladder polyp (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic cyst (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 2 (2) | 1 (1)
Hepatic steatosis (Hepatobiliary disorders) | 3 (3) | 1 (1)
Hepatomegaly (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hyperplastic cholecystopathy (Hepatobiliary disorders) | 2 (2) | 0 (0)
Non-alcoholic fatty liver (Hepatobiliary disorders) | 4 (4) | 3 (3)
Non-alcoholic steatohepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Post cholecystectomy syndrome (Hepatobiliary disorders) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0)
Food allergy (Immune system disorders) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 3 (3) | 1 (1)
Acute sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Bacterial infection (Infections and infestations) | 1 (2) | 1 (1)
Body tinea (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 2 (2) | 2 (2)
Candida infection (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1)
Conjunctivitis (Infections and infestations) | 4 (4) | 2 (2)
Conjunctivitis bacterial (Infections and infestations) | 0 (0) | 2 (2)
Coronavirus infection (Infections and infestations) | 18 (18) | 8 (8)
Covid-19 (Infections and infestations) | 30 (30) | 16 (16)
Cystitis (Infections and infestations) | 6 (6) | 1 (1)
Dacryocystitis (Infections and infestations) | 1 (1) | 0 (0)
Dermatophytosis of nail (Infections and infestations) | 3 (3) | 1 (1)
Empyema (Infections and infestations) | 0 (0) | 1 (1)
Enteritis infectious (Infections and infestations) | 1 (1) | 0 (0)
Enterocolitis viral (Infections and infestations) | 1 (1) | 1 (1)
Exanthema subitum (Infections and infestations) | 0 (0) | 1 (1)
Folliculitis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 5 (5) | 5 (6)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1)
Gingivitis (Infections and infestations) | 2 (2) | 1 (1)
Helicobacter gastritis (Infections and infestations) | 1 (1) | 0 (0)
Helicobacter infection (Infections and infestations) | 1 (1) | 0 (0)
Hepatitis e (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 7 (7) | 4 (4)
Hordeolum (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 1 (1)
Nasal herpes (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 22 (32) | 17 (20)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0)
Otitis externa (Infections and infestations) | 3 (3) | 1 (1)
Otitis media (Infections and infestations) | 1 (1) | 0 (0)
Periodontitis (Infections and infestations) | 3 (3) | 4 (4)
Pharyngitis (Infections and infestations) | 5 (8) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Post-acute covid-19 syndrome (Infections and infestations) | 1 (1) | 1 (1)
Rhinitis (Infections and infestations) | 1 (1) | 1 (1)
Skin bacterial infection (Infections and infestations) | 1 (1) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0)
Tinea pedis (Infections and infestations) | 2 (2) | 0 (0)
Tonsillitis (Infections and infestations) | 3 (4) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Vulvitis (Infections and infestations) | 1/113 (1) | 0/53 (0)
Vulvovaginal candidiasis (Infections and infestations) | 2/113 (2) | 0/53 (0)
Animal bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arthropod sting (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Avulsion fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Bone contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Chillblains (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 3 (5) | 5 (5)
Face injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fractured coccyx (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Gingival injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Heat illness (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Immunisation reaction (Injury, poisoning and procedural complications) | 7 (8) | 2 (4)
Inflammation of wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Nasal injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Neck injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Tooth fracture (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Vaccination complication (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 6 (6) | 0 (0)
Amylase increased (Investigations) | 3 (3) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 5 (5) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 0 (0)
Blood triglycerides increased (Investigations) | 1 (1) | 0 (0)
Carcinoembryonic antigen increased (Investigations) | 0 (0) | 1 (1)
Diagnostic aspiration (Investigations) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 3 (3) | 0 (0)
Helicobacter test positive (Investigations) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 12 (12) | 1 (1)
Occult blood positive (Investigations) | 1 (1) | 0 (0)
Pancreatic enzymes increased (Investigations) | 2 (2) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 16 (16) | 6 (6)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Dyslipidaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 7 (10) | 8 (9)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperlipasaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Zinc deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (9) | 8 (8)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 12 (13) | 4 (4)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (5) | 4 (5)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Nodal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 6 (7) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2)
Periarthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal ligament ossification (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Trigger finger (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastrointestinal submucosal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/278 (1) | 0/142 (0)
Pyogenic granuloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2/113 (2) | 0/53 (0)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Cervical radiculopathy (Nervous system disorders) | 3 (3) | 0 (0)
Diabetic neuropathy (Nervous system disorders) | 4 (4) | 0 (0)
Dizziness (Nervous system disorders) | 6 (6) | 5 (5)
Dizziness postural (Nervous system disorders) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0)
Head discomfort (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 12 (12) | 8 (11)
Hypoaesthesia (Nervous system disorders) | 6 (6) | 0 (0)
Intercostal neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Post herpetic neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Taste disorder (Nervous system disorders) | 2 (2) | 0 (0)
Tension headache (Nervous system disorders) | 0 (0) | 1 (1)
Anxiety disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Depressive symptom (Psychiatric disorders) | 1 (1) | 0 (0)
Initial insomnia (Psychiatric disorders) | 1 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 2 (3)
Sleep disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Calculus urethral (Renal and urinary disorders) | 1 (1) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 1 (1) | 0 (0)
Diabetic nephropathy (Renal and urinary disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 3 (3) | 0 (0)
Hypertonic bladder (Renal and urinary disorders) | 3 (3) | 0 (0)
Renal cyst (Renal and urinary disorders) | 3 (3) | 3 (3)
Ureterolithiasis (Renal and urinary disorders) | 2 (2) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Amenorrhoea (Reproductive system and breast disorders) | 1/113 (1) | 0/53 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1/278 (1) | 1/142 (1)
Endometrial disorder (Reproductive system and breast disorders) | 1/113 (1) | 0/53 (0)
Endometriosis (Reproductive system and breast disorders) | 1/113 (1) | 0/53 (0)
Intermenstrual bleeding (Reproductive system and breast disorders) | 0/113 (0) | 1/53 (1)
Menopausal symptoms (Reproductive system and breast disorders) | 1/113 (1) | 0/53 (0)
Pelvic cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 1/278 (1) | 0/142 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Cough variant asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Vasomotor rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Androgenetic alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1)
Dermatosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Dyshidrotic eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 3 (3) | 6 (6)
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Hand dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Miliaria (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Palmoplantar keratoderma (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (3)
Urticaria (Skin and subcutaneous tissue disorders) | 5 (7) | 1 (1)
Breast conserving surgery (Surgical and medical procedures) | 0 (0) | 1 (1)
Cataract operation (Surgical and medical procedures) | 5 (6) | 0 (0)
Cervical conisation (Surgical and medical procedures) | 1/113 (1) | 0/53 (0)
Coronary arterial stent insertion (Surgical and medical procedures) | 1 (1) | 0 (0)
Internal fixation of fracture (Surgical and medical procedures) | 1 (1) | 0 (0)
Intraocular lens implant (Surgical and medical procedures) | 2 (3) | 2 (3)
Large intestinal polypectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Lipoma excision (Surgical and medical procedures) | 0 (0) | 1 (1)
Medical device removal (Surgical and medical procedures) | 1 (1) | 0 (0)
Meniscus removal (Surgical and medical procedures) | 0 (0) | 1 (1)
Nephrectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Polypectomy (Surgical and medical procedures) | 2 (2) | 0 (0)
Rectal polypectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Synovial cyst removal (Surgical and medical procedures) | 1 (1) | 0 (0)
Tooth extraction (Surgical and medical procedures) | 3 (3) | 3 (3)
Tumour excision (Surgical and medical procedures) | 1 (1) | 0 (0)
Arteriosclerosis (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 10 (10) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Internal haemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0)
Raynaud's phenomenon (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-12-15): https://cdn.clinicaltrials.gov/large-docs/20/NCT04809220/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-14): https://cdn.clinicaltrials.gov/large-docs/20/NCT04809220/SAP_001.pdf